CLINICAL TRIAL: NCT00949273
Title: A Randomized, Controlled, Multicenter Trial to Evaluate the Safety and Efficacy of Cylindrical Abdominoperineal Resection in the Treatment of Advanced Very Low Rectal Cancer
Brief Title: Safety and Efficacy Study of Cylindrical Abdominoperineal Resection to Treat Rectal Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Chao Yang Hospital (Other)
Collaborators: Shandong Provincial Hospital (Other Government); Shandong Cancer Hospital and Institute (Other); The First Affiliated Hospital of Zhengzhou University (Other); Wuhan University (Other); Shenyang Anorectal Hospital (Other); Beijing Luhe Hospital (Other)
Responsible Party: Principal Investigator, Zhen Jun Wang, Professor and Head of General Surgery, Beijing Chao Yang Hospital
Other Study IDs: CAPR0668
Record Dates: First submitted 2009-07-29; First posted 2009-07-30 (Estimated); Last update posted 2013-11-28 (Estimated); Status verified 2013-11

CONDITIONS: Rectal Cancer; Treatment; Postoperative Complications; Neoplasm Recurrence, Local; Survival Rate
Keywords: cylindrical abdominoperineal resection; rectal cancer; acellular dermal matrix; pelvic reconstruction; circumferential resection margin; overall survival
MeSH Terms: conditions — Rectal Neoplasms; Postoperative Complications; Neoplasm Recurrence, Local

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — circumferential resection margin; bowel perforation; cross sectional tissue area outside the internal sphincter; mean distance from the internal sphincter to the anterior, posterior and lateral circumferential resection margins
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- cylindrical abdominoperineal resection: patients underwent cylindrical abdominoperineal resection for advanced very low rectal cancer
  Interventions: Procedure: cylindrical abdominoperineal resection
- abdominoperineal resection: patients underwent conventional abdominoperineal resection for advanced very low rectal cancer

INTERVENTIONS:
Procedure: cylindrical abdominoperineal resection — Extended abdominoperineal resection with human acellular dermal matrix reconstruction of the pelvic floor for rectal cancer
  Other Names: Ruinuo
  Groups: cylindrical abdominoperineal resection

SUMMARY:
The purpose of this study is to determine whether cylindrical abdominoperineal resection is effective in the treatment of advanced very low rectal cancer

DETAILED DESCRIPTION:
Abdominoperineal resection (APR) is still a common operation in patients with tumours less than 6 cm from the anal verge. The perineal phase of APR is a difficult part of the operation, often done with the patient in the supine position.The risk of inadvertent bowel perforation is high, the resulting specimen frequently has a waist at the lower border of the mesorectum, and the circumferential resection margin (CRM) is often close to the rectal muscle tube. The cylindrical APR may be performed via an extended posterior perineal approach, that aims to create a more cylindrical specimen without a waist. The potential benefit of this technique is a reduction in the risk of bowel perforation and tumour involvement of the CRM, and thus in the risk of local recurrence.

Perineal wounds in patients following APR are at considerable risk for infection, dehiscence and delayed healing when closed primarily. This can be further increased in patients who have received neoadjuvant chemoradiation therapy. The adoption of extended resection, such as the cylindrical APR, may cause additional risks. The use of acellular biomaterials, including human acellular dermal matrix (HADM) has drawn great interest for the complex abdominal wall reconstruction.

The purpose of this study is to determine whether cylindrical abdominoperineal resection is effective in the treatment of advanced very low rectal cancer, and to determine the initial results of pelvic reconstruction using human acellular dermal matrix after cylindrical abdominoperineal resection.

ELIGIBILITY:
Inclusion Criteria:

* Tumor within 6 cm of the anal verge, or with very narrow pelvis
* T3-T4 as determined by preoperative MRI or endorectal ultrasonography examination, or a low tumor is fixed or tethered at rectal examination
* Absence of distant metastases
* Absence of intestinal obstruction

Exclusion Criteria:

* T1-T2 as determined by preoperative MRI or endorectal ultrasonography examination
* with distant metastases
* with intestinal obstruction
* pregnancy or lactation
* allergic constitution to heterogeneous protein
* with operation contraindication
* with mental disorder

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: hospitalized patients with rectal cancer
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2009-07; Primary Completion 2013-11 (Estimated); Study Completion 2013-11 (Estimated)

PRIMARY OUTCOMES:
postoperative complications | 08/01/2011

SECONDARY OUTCOMES:
3-years overall survival | 08/01/2013

CONTACTS AND LOCATIONS:
Overall Officials: Zhen Jun Wang, M.D., Study Chair — Beijing Chao Yang Hospital; Yong Dai, M.D., Principal Investigator — Shandong Provincial Hospital; Heng Ma, M.D., Principal Investigator — Shandong Cancer Hospital and Institute; Qun Qian, M.D., Principal Investigator — Zhong Nan Hospital, Wuhan University; Xian Dong Zeng, M.D., Principal Investigator — Shenyang Anorectal Hospital; Jian Hua Cai, M.D., Principal Investigator — Beijing Luhe Hospital; Wei Tang Yuan, M.D., Principal Investigator — The First Affiliated Hospital of Zhengzhou University
Locations (7):
- China (7):
  - Beijing Luhe Hospital, Beijing, Beijing Municipality
  - General Surgery, Beijing Chao Yang Hospital, Beijing, Beijing Municipality
  - The first Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Zhongnan Hospital, Wuhan University, Wuhan, Hubei
  - Shenyang Anorectal Hospital, Shenyang, Liaoning
  - General Surgery, Shandong Provincial Hospital, Jinan, Shandong
  - Shandong Cancer Hospital and Institute, Jinan, Shandong

REFERENCES:
- [Result] Holm T, Ljung A, Haggmark T, Jurell G, Lagergren J. Extended abdominoperineal resection with gluteus maximus flap reconstruction of the pelvic floor for rectal cancer. Br J Surg. 2007 Feb;94(2):232-8. doi: 10.1002/bjs.5489. PMID 17143848